CLINICAL TRIAL: NCT06830499
Title: Safety, Effectiveness and Durability of Sapien 3 Transcatheter Aortic Valve Replacement in Young Aortic Valve Stenosis Patients From China
Brief Title: Sapien 3 Transcatheter Aortic Valve Replacement in Young Aortic Valve Stenosis Patients From China
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Fu Wai Hospital, Beijing, China (Other); West China Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: China Young TAVR Study
Record Dates: First submitted 2025-01-09; First posted 2025-02-17 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-01

CONDITIONS: AORTIC VALVE DISEASES; Bicuspid Aortic Valve (BAV)
Keywords: TAVR; real-world; aortic valve stenosis; Sapien 3
MeSH Terms: conditions — Aortic Valve Disease; Bicuspid Aortic Valve Disease; Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 300 retrospectively enrolled patients: Procedure: TAVR
  Interventions: Procedure: Transcatheter Aortic Valve Replacement (TAVR)
- 150 prospectively enrolled patients: Procedure: TAVR
  Interventions: Procedure: Transcatheter Aortic Valve Replacement (TAVR)

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Replacement (TAVR) — TAVR procedure was performed according to standard clinical practice. Successful vascular access, delivery and deployment of the device and successful retrieval of the delivery system will be attempted. Vascular access site will be through transfemoral on the basis of pre-procedural evaluation of access site vessel. The procedure will be performed under local or general anesthesia and per clinical practice standard.

SUMMARY:
Safety, effectiveness and durability of Sapien 3 transcatheter aortic valve replacement in young aortic valve stenosis patients from China：A multi-center, retrospective and prospective, single arm, observational study

DETAILED DESCRIPTION:
Transcatheter aortic valve replacement (TAVR) has revolutionized the treatment of patients with severe aortic stenosis (AS). Currently TAVR indication has expanded to intermediate and low-risk patients from inoperable or high-risk patients, through a rigorous series of clinical trials comparing TAVR with surgical aortic valve replacement (SAVR).

Despite 2020 American College of Cardiology (ACC)/American Heart Association (AHA) guidelines recommended SAVR for patients with symptomatic severe AS aged <65 years, the previous data from United States nationwide Vizient Clinical Data Base and Northern New England Cardiovascular Disease Group Consortium (NNECDSG) registry demonstrated dramatic growth in TAVR utilization in younger patients aged <65 years from 2015 to 2021/2022, which is possibly driven by increased TAVR utilization in low surgical risk patients.

However, TAVR has never been systematically tested in young (<65 years old), low-risk patients, with many unanswered questions, especially the safety and effectiveness of TAVR in patients with bicuspid aortic valves and the durability of transcatheter heart valves. Furthermore, we noticed that the patients between 65 years old and 70 years old accounted for 23.3% of all the TAVR patients and this patient subgroup were underrepresented in the previous study, which makes it necessary to also explore the interested endpoints in this subgroup.

The aim of this study is to establish the safety and efficacy of Sapien 3 TAVR in young (50~70 years old) Chinese patients with severe symptomatic AS, including Type-1 bicuspid population and to explore the durability performance of Sapien 3 in this cohort.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL of the following inclusion criteria to be eligible for participation:

* 50 years of age or older but ≤70 years old at time of consent.
* Severe AS, defined as follows:

  a) For symptomatic patients: i) Aortic valve area ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), OR mean gradient ≥40 mm Hg, OR Maximal aortic valve velocity ≥4.0 m/sec by transthoracic echocardiography at rest b) For asymptomatic patients: i) Very severe AS with an aortic valve area of ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), AND maximal aortic velocity ≥5.0 m/sec, or mean gradient ≥60 mm Hg by transthoracic echocardiography at rest, OR ii) Aortic valve area of ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), AND a mean gradient ≥40 mm Hg or maximal aortic valve velocity ≥4.0 m/sec by transthoracic echocardiography at rest, AND an exercise tolerance test that demonstrates a limited exercise capacity, abnormal BP response, or arrhythmia OR iii) Aortic valve area of ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), AND mean gradient ≥40 mmHg, or maximal aortic valve velocity ≥4.0 m/sec by transthoracic echocardiography at rest, AND a left ventricular ejection fraction <50%.
* Tricuspid aortic valve stenosis and type-1 bicuspid aortic valve anatomy confirmed by MDCT.
* The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.
* Adequate iliofemoral access and acceptable level of vessel calcification and tortuosity for safe device implant.
* The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.

Exclusion Criteria:

Subjects are NOT eligible for participation if they meet ANY of the following exclusion criteria:

* Any of the following: a. no calcification; b. challenging calcification based on physician's experience and discretion (Case Review Board would decide whether to exclude challenging calcification cases).
* Aortic valve is a congenital unicuspid valve, congenital Type-0 or Type-2 bicuspid valve, or quadricuspid valve.
* Severe femoral, iliac or aortic atherosclerosis, calcification, coarctation, aneurysm or tortuosity, which prevents transfemoral TAVR.
* Evidence of an acute myocardial infarction ≤ 1 month (30 days), with evidence of myocardial necrosis in a clinical setting consistent with acute myocardial ischemia.
* Need for open heart surgery (including severe aortic regurgitation, mitral regurgitation or stenosis, or tricuspid regurgitation, congenital heart disease, AF, complex coronary artery disease).
* Aortic disease: a. bicuspid aortic valve with an ascending aorta diameter ≥ 45mm b. tricuspid aortic valve with an ascending aorta diameter ≥ 50mm.
* Pre-existing mechanical or bioprosthetic valve in any position.
* Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of the screening visit.
* Emergency interventional/surgical procedures within 30 days of the valve implant procedure.
* Hypertrophic cardiomyopathy with or without obstruction.
* Ventricular dysfunction with LVEF < 30%.
* Cardiac imaging (echo, CT, and/or MRI) evidence of ventricular mass, thrombus or vegetation.
* Inability (including allergy) to heparin, iodine contrast agent, warfarin or NOAC, aspirin or clopidogrel.
* Stroke or transient ischemic attack (TIA) within 180 days of the valve implant procedure.
* Renal replacement therapy at the time of screening.
* Severe lung disease (FEV1 < 50% predicted) or currently on home oxygen.
* Estimated life expectancy < 24 months.
* Currently participating in an investigational drug or another device study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials. Observational studies are not considered exclusionary.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Young (50~70 years old) Chinese patients with severe symptomatic AS, including Type-1 bicuspid population
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | At 5 years
  The primary end point is the 5 year all-cause mortality

SECONDARY OUTCOMES:
The composite of all-cause mortality, stroke and rehospitalization | At 30 days, 1, 3, 5 years
  The composite of all-cause mortality, stroke, rehospitalization (procedure, valve and heart failure related) at 30 days, 1, 3, 5 years
The composite of device success | At 30 days
  The composite of device success at 30 days comprising the following: freedom from mortality, successful access, delivery of the device, and retrieval of the delivery system, correct positioning of a single prosthetic heart valve into the proper anatomical location, freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication, intended performance of the valve (mean gradient <20 mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation), according to the VARC-3 definition
The durability performance of Sapien 3 | At 1, 3, 5 years
  The durability performance of Sapien 3 at 1, 3, 5 years: bioprosthetic valve dysfunction (BVD, including SVD, non-SVD, endocarditis and thrombosis), moderate or severe hemodynamic valve deterioration (HVD), bioprosthetic valve failure (BVF) according to the VARC-3 definition, EOA/mean gradient (MG) change over follow up
Annular rupture | At 1 day of discharge
  The incidence of annular rupture
Paravalvular leakage | At 1 day of discharge, 30 days, 1, 3, 5 years
  The incidence of paravalvular leakage
Technical success | At exit from procedure room
  Technical success (at exit from procedure room):
  * freedom from mortality
  * successful access, delivery of the device, and retrieval of the delivery system
  * correct positioning of a single prosthetic heart valve into the proper anatomical location
  * freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
Procedural success | At 30 days
  Procedural success at 30 days defined as meeting all of the following:
  * Device success
  * No device or procedure related SAE's as follows:
    1. Life-threatening bleed (BARC 3b or greater)
    2. Major vascular or cardiac structural complications requiring unplanned reintervention or surgery
    3. Stage 2 or 3 AKI (includes new dialysis)
    4. MI or need for PCI/CABG
    5. Severe heart failure or hypotension requiring IV inotrope >12 hours, ultrafiltration or mechanical circulatory support
    6. Prolonged intubation > 48 hours
    7. Need for a permanent pacemaker implant or continuous, new onset atrial fibrillation
Mortality (all cause & cardiovascular) | At 30 days, 1, 3, 5 years
  The incidence of mortality (all cause & cardiovascular)
Stroke (disabling and nondisabling) | At 30 days, 1, 3, 5 years
  The incidence of stroke (disabling and nondisabling)
Rehospitalization (procedure, valve and heart failure related) | At 30 days, 1, 3, 5 years
  The incidence of rehospitalization (procedure, valve and heart failure related)
Major vascular complication | At 30 days, 1, 3, 5 years
  The incidence of major vascular complication
Major or life-threatening bleeding | At 30 days, 1, 3, 5 years
  The incidence of major or life-threatening bleeding
Myocardial infarction | At 30 days, 1, 3, 5 years
  The incidence of myocardial infarction
Acute kidney injury stage 2 or 3 | At 30 days, 1, 3, 5 years
  The incidence of acute kidney injury stage 2 or 3
Need for a permanent pacemaker | At 30 days, 1, 3, 5 years
  The incidence of permanent pacemaker implantation
New onset atrial fibrillation | At 30 days, 1, 3, 5 years
  The incidence of new onset atrial fibrillation
Valve endocarditis | At 30 days, 1, 3, 5 years
  The incidence of valve endocarditis
Valve thrombosis | At 30 days, 1, 3, 5 years
  The incidence of valve thrombosis
New York Heart Association class | At 30 days, 1, 3, 5 years
  The changes in New York Heart Association class
Patient-prosthesis mismatch | At 30 days, 1, 3, 5 years
  The incidence of patient-prosthesis mismatch
Health status as evaluated by Quality of Life questionnaires - KCCQ | At baseline, 30 days, 1, 3, 5 years
  The changes in Health status as evaluated by Quality of Life questionnaires - KCCQ

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yang, MD, PhD, Principal Investigator — Department of Cardiovascular Surgery of Xijing Hospital, Air Force Military Medical University
Locations (4):
- China (4):
  - Department of Cardiovascular Surgery of Xijing Hospital, Air Force Military Medical University, Xi'an, Shaanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing
  - Shanghai Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) would not be shared, according to local authority data privacy policy.

REFERENCES:
- [Background] Ten Berg J, Sibbing D, Rocca B, Van Belle E, Chevalier B, Collet JP, Dudek D, Gilard M, Gorog DA, Grapsa J, Grove EL, Lancellotti P, Petronio AS, Rubboli A, Torracca L, Vilahur G, Witkowski A, Mehilli J. Management of antithrombotic therapy in patients undergoing transcatheter aortic valve implantation: a consensus document of the ESC Working Group on Thrombosis and the European Association of Percutaneous Cardiovascular Interventions (EAPCI), in collaboration with the ESC Council on Valvular Heart Disease. Eur Heart J. 2021 Jun 14;42(23):2265-2269. doi: 10.1093/eurheartj/ehab196. PMID 33822924
- [Background] Gupta T, DeVries JT, Gilani F, Hassan A, Ross CS, Dauerman HL. Temporal Trends in Transcatheter Aortic Valve Replacement for Isolated Severe Aortic Stenosis. J Soc Cardiovasc Angiogr Interv. 2024 Apr 5;3(7):101861. doi: 10.1016/j.jscai.2024.101861. eCollection 2024 Jul. No abstract available. PMID 39132009
- [Background] Sharma T, Krishnan AM, Lahoud R, Polomsky M, Dauerman HL. National Trends in TAVR and SAVR for Patients With Severe Isolated Aortic Stenosis. J Am Coll Cardiol. 2022 Nov 22;80(21):2054-2056. doi: 10.1016/j.jacc.2022.08.787. Epub 2022 Sep 16. No abstract available. PMID 36122626
- [Background] Popma JJ, Deeb GM, Yakubov SJ, Mumtaz M, Gada H, O'Hair D, Bajwa T, Heiser JC, Merhi W, Kleiman NS, Askew J, Sorajja P, Rovin J, Chetcuti SJ, Adams DH, Teirstein PS, Zorn GL 3rd, Forrest JK, Tchetche D, Resar J, Walton A, Piazza N, Ramlawi B, Robinson N, Petrossian G, Gleason TG, Oh JK, Boulware MJ, Qiao H, Mugglin AS, Reardon MJ; Evolut Low Risk Trial Investigators. Transcatheter Aortic-Valve Replacement with a Self-Expanding Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1706-1715. doi: 10.1056/NEJMoa1816885. Epub 2019 Mar 16. PMID 30883053
- [Background] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Background] Reardon MJ, Van Mieghem NM, Popma JJ, Kleiman NS, Sondergaard L, Mumtaz M, Adams DH, Deeb GM, Maini B, Gada H, Chetcuti S, Gleason T, Heiser J, Lange R, Merhi W, Oh JK, Olsen PS, Piazza N, Williams M, Windecker S, Yakubov SJ, Grube E, Makkar R, Lee JS, Conte J, Vang E, Nguyen H, Chang Y, Mugglin AS, Serruys PW, Kappetein AP; SURTAVI Investigators. Surgical or Transcatheter Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2017 Apr 6;376(14):1321-1331. doi: 10.1056/NEJMoa1700456. Epub 2017 Mar 17. PMID 28304219
- [Background] Leon MB, Smith CR, Mack MJ, Makkar RR, Svensson LG, Kodali SK, Thourani VH, Tuzcu EM, Miller DC, Herrmann HC, Doshi D, Cohen DJ, Pichard AD, Kapadia S, Dewey T, Babaliaros V, Szeto WY, Williams MR, Kereiakes D, Zajarias A, Greason KL, Whisenant BK, Hodson RW, Moses JW, Trento A, Brown DL, Fearon WF, Pibarot P, Hahn RT, Jaber WA, Anderson WN, Alu MC, Webb JG; PARTNER 2 Investigators. Transcatheter or Surgical Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2016 Apr 28;374(17):1609-20. doi: 10.1056/NEJMoa1514616. Epub 2016 Apr 2. PMID 27040324
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243